CLINICAL TRIAL: NCT04879342
Title: Evaluation of Values in Perspective (VIP) Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Marie Guerda Nicolas, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20201386
Record Dates: First submitted 2021-05-04; First posted 2021-05-10 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Risk Behavior
MeSH Terms: conditions — Risk-Taking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VIP Program Group (Experimental): Participants in this group will receive a 26 week course on risk reduction strategies.
  Interventions: Behavioral: VIP Program

INTERVENTIONS:
Behavioral: VIP Program — This intervention will engage the participants with psychoeducational material once a week. This material will include didactic instruction as well as participant engagement in developmentally appropriate activities.

SUMMARY:
The primary purpose of this study is to evaluate the effectiveness and perceived usefulness of the Values in Perspective (VIP) program in reducing and preventing engagement in risky behaviors among youths. The VIP program is a structured, values-based intervention designed to promote self-awareness, ethical decision-making, and long-term goal setting in young people. This study aims to assess how participation in the program influences youths' attitudes, knowledge, and behaviors related to common adolescent risk factors such as substance use, unsafe sexual activity, and delinquency. The goal is to determine whether the VIP program can serve as a scalable and culturally relevant prevention strategy to promote positive youth development and reduce high-risk behaviors in middle and high school-aged youths.

ELIGIBILITY:
Inclusion criteria

1. A youth residing in Miami-Dade County.
2. Must be in grades 6-12 and must be eligible for free and reduced lunch.
3. Must be able to speak and read English proficiently.

Exclusion criteria

1. Does not reside in Miami-Dade County.
2. Does not comprehend, speak, or read English proficiently.
3. In elementary school.
4. In high-income household as evidenced by not qualifying for free and reduced lunch.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 850 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
SRAE Scores - Middle School | Up to 26 weeks
  Sexual Risk Avoidance Education Program (SRAE) for middle school participants has a total score ranging from 0 to 170 with a higher score indicating higher risk behavior.
SRAE Scores - High School | Up to 26 weeks
  Sexual Risk Avoidance Education Program (SRAE) for high school participants has a total score ranging from 0 to 190 with a higher score indicating higher risk behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Guerda Nicolas, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No